CLINICAL TRIAL: NCT05180890
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, 3-Period Crossover Study to Evaluate the Safety, Tolerability, Pharmacodynamic, and Pharmacokinetic Effects of Overnight Intravenous TAK-925 in Patients With Obstructive Sleep Apnea
Brief Title: A Study of Danavorexton (TAK-925) in Adults With Obstructive Sleep Apnea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TAK-925-1020
Record Dates: First submitted 2022-01-03; First posted 2022-01-06 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Sleep Apnea
Keywords: Drug Therapy
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — TAK-925

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo infusion, intravenously, administered overnight for approximately 10-hours on Days 1 to 2 in each Treatment Period 1, 2, or 3.
  Interventions: Drug: Placebo
- Danavorexton LD (Experimental): Danavorexton LD regimen, infusion, intravenously, administered overnight for approximately 10-hours on Days 1 to 2 in each Treatment Period 1, 2, or 3.
  Interventions: Drug: Danavorexton
- Danavorexton HD (Experimental): Danavorexton HD regimen, infusion, intravenously, administered overnight for approximately 10-hours on Days 1 to 2 in each Treatment Period 1, 2, or 3.
  Interventions: Drug: Danavorexton

INTERVENTIONS:
Drug: Danavorexton — Danavorexton intravenous infusion.
  Other Names: TAK-925
  Arms: Danavorexton HD; Danavorexton LD
Drug: Placebo — Placebo intravenous infusion.
  Arms: Placebo

SUMMARY:
The main aim of the study is to check the side effects from overnight treatment with danavorexton and assess the tolerability of varying doses of danavorexton administered intravenously.

Before starting treatment with danavorexton, participants will keep a sleep diary and use an under-mattress sensor for at least 7 nights to check regular sleep habits.

There will be 3 Treatment Period up to 14 days apart. In each Treatment Period, participants will receive an intravenous (through the vein) infusion of either danavorexton or a placebo starting in the evening and continuing over a 10-hour period. A placebo looks exactly like danavorexton but does not have any medicine in it.

Participants will take part in a follow-up phone appointment about a week after the last Treatment Period.

DETAILED DESCRIPTION:
The drug being tested in this study is called danavorexton. The study will look at the safety, tolerability, pharmacokinetic (PK), and pharmacodynamics (PD) effects of danavorexton.

The study will enroll approximately 18 participants (to acquire data in 'n' greater than or equal to [>=] 12). Each participant will receive one of the following treatments in each Treatment Period: Danavorexton low dose (LD), danavorexton high dose (HD), or placebo. All participants will receive all 3 treatments. A washout period of a minimum of 2 days up to 14 days will be maintained between the end of infusion to the start time of next infusion. The order in which each participant receives the 3 treatments will be randomly assigned. Treatment order will remain undisclosed to the participants and study doctor during the study (unless there is an urgent medical need).

This single-center trial will be conducted in Australia. The overall time to participate in this study is up to 69 days. Participants will be followed remotely until 5 to 9 days after the last dose of study drug in the Treatment Period 3.

ELIGIBILITY:
Inclusion Criteria:

1. Has OSA diagnosed according to the International Classification of Sleep Disorders-3 (ICSD-3) criteria and an AHI of 12-50 events/hour sleep (documented by an in-clinic PSG or at-home sleep test within the last 12 months). Participants who do not have PSG results from within 12 months available may be offered a screening home sleep test.
2. Those who use continuous positive airway pressure (CPAP), oral appliance, or hypoglossal nerve stimulator must be willing to forego this therapy during all in-clinic PSGs and during the home sleep test if one is required.
3. Has no known history of a sleep disorder other than OSA based on interviews at the screening visit, such as, for example, restless legs syndrome accompanied by periodic leg movements of sleep.
4. Has a regular bedtime (example, between 8 p.m. - 1 a.m.) and regular time in bed averaging between 6.0 and 10.0 hours/night, as verified by sleep tracking mat and sleep diary data. Sleep durations and bedtimes outside of this range can be discussed for inclusion on a case by case basis with the sponsor.
5. Has a body mass index (BMI) of 18 to 38.5 kilogram per square meter (kg/m^2) inclusive.

Exclusion Criteria:

1. Has an occupation requiring nighttime shift work or variable shift work within the past 2 months or has travelled with significant jet lag within 14 days before the study start or plans to travel with significant jet lag during the study.
2. Has nicotine dependence that is likely to have an effect on sleep (example, a participant who routinely awakens at night to smoke) or challenge the conduct of this study (smokes >=10 cigarettes/day), or the participant is unwilling to discontinue all smoking and nicotine use during the confinement periods.
3. Has a caffeine consumption of more than 600 milligram (mg)/day for 7 days before Period 1 Day 1 (1 serving of coffee is approximately equivalent to 120 mg of caffeine; 16 ounces of cola or energy drink contain approximately 39 and 148 mg of caffeine, respectively).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants With at Least one Treatment-emergent Adverse Event (TEAE) | From the first dose of danavorexton in Treatment Period 1 up to approximately 7 days after the last dose of danavorexton in Treatment Period 3 (up to 41 days)

SECONDARY OUTCOMES:
Change From Baseline in Upper Airway Collapsibility Index (UACI) | Baseline (-15 minutes from the start of infusion [first UACI]), and at 20 minutes (second UACI), and 55 minutes (third UACI) on Day 1 of each Treatment Period
  The UACI is a 10-minute evaluation that tests the key biological mechanism that causes obstructive sleep apnea (OSA).
Apnea-Hypopnea Index (AHI) Observed During Overnight Polysomnographys (PSGs) | Day 1 up to Day 2 of each Treatment Period
  PSG analysis will be performed to determine an apnea hypopnea index. AHI score is used to indicate the severity of sleep apnea. The AHI is calculated by dividing the number of apnea events by the number of hours of sleep. An apnea hypopnea index less than five events per hour is considered within normal limits.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Adelaide Institute for Sleep Health (AISH), Flinders University, Adelaide, Australia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click on this link — https://clinicaltrials.takeda.com/study-detail/5af25efdcb954c82?idFilter=%5B%22TAK-925-1020%22%5D